CLINICAL TRIAL: NCT02837237
Title: A Phase 1, Open-Label Study in Hemodialysis and Non-Hemodialysis Patients With Severe Chronic Kidney Disease to Evaluate the Safety, Tolerability, and Pharmacokinetics of KBP-5074 Following Oral Administration
Brief Title: Safety, Tolerability, and Pharmacokinetics of KBP-5074 Following Oral Administration in Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KBP Biosciences (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KBP5074-1-003
Record Dates: First submitted 2016-07-11; First posted 2016-07-19 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — KBP-5074

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KBP-5074 (Experimental): Single oral dose
  Interventions: Drug: KBP-5074

INTERVENTIONS:
Drug: KBP-5074 — In Part 1 of the study, non-HD patients with severe CKD in Cohort 1 will receive a single oral capsule dose of KBP-5074 on Day 1 following a fast between 2 and 4 hours.
  In Part 2 of the study, HD patients with severe CKD will receive a single oral capsule dose of KBP-5074 following a fast between 2 and 4 hours. The dose of KBP 5074 will be administered on Day 1 immediately following a dialysis session.
  Other Names: KBP-5074 mineralocorticoid receptor antagonist

SUMMARY:
This study explores the use of KBP-5074 in patients with advanced stages of Chronic Kidney Disease (CKD) (including patients with severe renal impairment and those on hemodialysis [HD]) and to assess the safety, tolerability, and pharmacokinetics (PK) of single doses of KBP-5074 in male and female patients with severe CKD (defined as estimated glomerular filtration rate [eGFR] ≥15 mL/min/1.73 m2 and ≤29 mL/min/1.73 m2, based on the Modification of Diet in Renal Disease [MDRD] equation) and a subset of patients requiring HD.

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label, 2-part study designed to assess the PK, safety, and tolerability of KBP-5074 in patients undergoing HD and non-HD patients with severe CKD (defined using the eGFR ≥15 mL/min/1.73 m2 and ≤29 mL/min/1.73 m2 based on the MDRD equation). The study will be conducted at up to 4 clinical research units (CRUs) in the US. Approximately 12 patients will be enrolled in the study (a single cohort of 6 patients in each of Part 1 and Part 2). Parts 1 and 2 of the study will be conducted in parallel. If Part 1 is completed prior to the completion of Part 2, or vice versa, the PK, safety, and tolerability analyses for the completed study part may proceed as planned and will not be delayed based on the timing of the other respective study part.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between 18 and 75 years of age, inclusive.
2. Body mass index (BMI) between 19 and 42 kg/m2, inclusive.
3. Has severe CKD, defined as eGFR ≥15 mL/min/1.73 m2 and ≤29 mL/min/1.73 m2 based on the IDMS traceable15 MDRD equation, according to laboratory results at Screening (non-HD patients only [Part 1]). Patients with a prior history of greater than 2 weeks of dialysis in the past and who have dialyzed in the 6 months prior to dosing on Day 1 will be excluded. Patients who have had temporary dialysis for acute kidney injury will be allowed at the discretion of the Investigator.
4. Serum potassium between 3.3 and 4.8 mmol/L, inclusive, at both Screening and Check-in (Day -1) (non-HD patients only [Part 1]). One repeat test will be allowed to exclude lab error or hemolyzed samples.
5. Is on a hemodialysis schedule for at least 45 days with KT/V ≥1.2 for end-stage renal disease (ESRD) regardless of the etiology including diabetes, with an average 3 hemodialysis sessions per week (HD patients only [Part 2]).
6. Is a nonsmoker or light smoker (smokes fewer than 10 cigarettes per day). Alcohol addressed in exclusion.
7. Female patients cannot be pregnant or lactating/breast-feeding and will either be postmenopausal (female patients who state they are postmenopausal should have had cessation of menses for >1 year and have serum follicle stimulating hormone [FSH] levels >40 mIU/mL and estradiol <20 pg/mL, surgically sterile (including bilateral tubal ligation, salpingectomy [with or without oophorectomy], surgical hysterectomy, or bilateral oophorectomy [with or without hysterectomy]) for at least 3 months prior to Screening, or will agree to use, from the time of Check-in (Day -1) until 90 days following the last dose of study drug, the following forms of contraception: double-barrier method, hormonal contraceptives, barrier with spermicide, diaphragm or cervical cap with spermicide, intrauterine device, oral, implantable, or injectable contraceptives, or a sterile sexual partner. All female patients will have a negative urine or serum pregnancy test result prior to enrollment in the study.
8. Male patients will either be surgically sterile or agree to use, from the time of Check-in (Day -1) until 90 days following the last dose of study drug, the following forms of contraception: male condom with spermicide and a female partner who is sterile or agrees to use hormonal contraceptives, female condom with spermicide, diaphragm or cervical cap with spermicide, intrauterine device, oral, implantable, or injectable contraceptives. Male patients will refrain from sperm donation from the time of Check-in (Day -1) until 90 days following the last dose of study drug.
9. Is capable of understanding the written informed consent, provides signed and witnessed written informed consent, and agrees to comply with protocol requirements.

Exclusion Criteria:

1. History of any prior or concomitant clinical condition or acute and/or unstable systemic disease compromising patient inclusion, at the discretion of the Investigator.
2. Has a history or presence of clinically significant (CS) cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease, which in the Investigator's opinion would not be suitable for the study from patient safety consideration and could interfere the results of the trial.
3. History of CS hypotension during the 6 months prior to the dose of study drug on Day 1 as determined by the Investigator.
4. History of symptomatic intradialytic hypotension as determined by the Investigator (mild to moderate decrease in blood pressure during dialysis is allowed; HD patients only [Part 2]).
5. History of CS hyperkalemia while on an angiotensin converting enzyme inhibitor, angiotensin receptor blocker, direct renin inhibitor, and/or MRA.
6. Hospitalization for hyperkalemia during the last 6 months prior to the dose of study drug on Day 1 or hyperkalemia >5.5 mmol/L during the 2 weeks prior to the Screening visit.
7. History of stroke within 3 months prior to the dose of study drug on Day 1.
8. History of cardiac transplant.
9. History of severe uncontrolled arrhythmia, acute myocardial infarction, or acute coronary syndrome within 3 months prior to the dose of study drug on Day 1.
10. Clinical diagnosis of heart failure and persistent symptoms (New York Heart Association Class II to IV) at either the Screening visit or at Check-in (Day 1).
11. History of stomach or intestinal surgery (except that cholecystectomy, appendectomy, and/or hernia repair will be allowed).
12. History of prescription drug abuse, illicit drug use, or alcohol abuse according to medical history within 6 months prior to the Screening visit or any alcohol use or for at least 48 hours prior to dosing on Day 1.
13. History of clinically significant acute or chronic hepatitis (including infectious, metabolic, autoimmune, genetic, ischemic, or other forms), hepatocirrhosis, or hepatic tumors.
14. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C (HCV) antibody. If a patient with Severe renal impairment or on HD has positive test results for HCV antibody but liver function tests are otherwise not CS, the patient may be included at the Investigator's discretion.
15. Clinically significant abnormal liver function test at screening or Check-in (Day -1), defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times upper limit of normal (ULN) or total bilirubin >ULN.
16. Recent (within 3 month prior to the dose of study drug on Day 1) or planned coronary revascularization by angioplasty or cardiovascular surgery (excluding HD vascular access).
17. Kidney transplant scheduled within the year.
18. Systolic blood pressure <90 or >200 mmHg and/or diastolic blood pressure <60 or >110 mmHg during the Screening visit and before the dose of study drug on Day 1; may be repeated at the discretion of the Investigator.
19. Positive screen for alcohol or drugs of abuse (except for patients with a positive drug screen test if it is a result of a prescribed medication from their physician) at Screening and Check-in (Day -1). Hemodialysis patients will be tested with serum drug screen at Screening and using salivary testing at Check-in (Day -1).
20. Female is pregnant or breastfeeding within 2 years prior to the dose of study drug on Day 1 or positive pregnancy test (serum/urine) result during the Screening visit and before the dose of study drug on Day 1. Patients who have a false positive test attributable to their post-menopausal state or kidney disease, as determined by the Investigator, will be allowed to participate.
21. Has a known hypersensitivity to KBP-5074, aldosterone antagonists, or related compounds.
22. Receipt of any other investigational product within 30 days or 5 half-lives (whichever is longer) prior to the dose of study drug on Day 1.
23. Currently on a MRA (eg, spironolactone, eplerenone) or potassium sparing diuretics (eg, amiloride, triamterene).
24. Concomitant use of or treatment with any prescription drugs, herbal products, vitamins, minerals, and over-the-counter medications within 14 days prior to Check in (Day -1) and during the study. Exceptions may be made on a case by case basis following discussion and agreement between the Investigator and the Sponsor. Patients requiring HD (Part 2) may continue to receive routine medications (including vitamins, antidepressants, antihypertensive, and low dose aspirin) to maintain their stable medication regimen.
25. Use of any nutrients known to modulate cytochrome P450 (CYP)3A activity (based on the KBP-5074 metabolic pathway) or any strong or moderate inhibitors or inducers of CYP3A4, starting from 14 days prior to dose administration on Day 1 until the final end of study assessments, including but not limited to the following: inhibitors such as ketoconazole, miconazole, itraconazole, fluconazole, atazanavir, erythromycin, clarithromycin, ranitidine, cimetidine, verapamil, and diltiazem and inducers such as rifampicin, rifabutin, glucocorticoids, carbamazepine, phenytoin, phenobarbital, and St. John's wort.
26. Participated in strenuous exercise from 48 hours prior to Check-in (Day -1) or during the study through the final end of study assessment.
27. Has donated or lost a significant volume (>500 mL) of blood or plasma within 30 days prior to Check-in (Day -1).
28. Is an employee or family member of the Investigator or study site personnel.
29. Has problems understanding the protocol requirements, instructions, study related restrictions, and/or problems understanding the nature, scope, and potential consequences of participating in this clinical study.
30. Is unlikely to comply with the protocol requirements, instructions, and/or study related restrictions (eg, uncooperative attitude, unavailable for follow up call, and/or improbability of completing the clinical study).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- KBP Biosciences USA Inc, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- KBP-5074: Single oral dose
  KBP-5074: In Part 1 of the study, non-HD patients with severe CKD in Cohort 1 will receive a single oral capsule dose of KBP-5074 on Day 1 following a fast between 2 and 4 hours.
  In Part 2 of the study, HD patients with severe CKD will receive a single oral capsule dose of KBP-5074 following a fast between 2 and 4 hours. The dose of KBP 5074 will be administered on Day 1 immediately following a dialysis session.
Period: Overall Study
Arm/Group | KBP-5074
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | KBP-5074
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 53.5 [37 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 124.8 (14.18)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events
Description: Physical exam, vital signs, EKG, clinical laboratory tests, adverse events
Time Frame: 312 hours
Measure: Count of Participants; unit: Participants
Arm/Group | KBP-5074
Number analyzed (Participants) | 11
Participants | 0

ADVERSE EVENTS:
Time Frame: 14 days
Description: An overall summary of the number and percentage of subjects in each category were presented, as well as an overall summary of the number of events in each category. The number and percentage of subjects reporting AEs in each category above were summarized by study part and cohort according to the system organ class (SOC) and preferred term (PT) assigned to the event using the Medical Dictionary for Regulatory Activities (MedDRA) version 19.0.
Arm/Group | KBP-5074
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 4/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KBP-5074 (N=11)
fatigue (General disorders) | 1 (1)
procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
increased creatinine (Investigations) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No